CLINICAL TRIAL: NCT05026021
Title: BKVIR Project: Predictive Biological Method of BKvirus Associated Nephropathy Risk by the NEPHROVIR Method
Brief Title: Prediction of BKvirus Nephropathy Risk by the NEPHROVIR Method in Kidney Transplant Patients With BKvirus Viremia
Acronym: BK-VIR
Status: Active, not recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: SATT Paris Saclay (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2020-A01443-36
Record Dates: First submitted 2021-06-07; First posted 2021-08-30 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-03

CONDITIONS: BK Virus Infection; Nephropathy; Kidney Transplantation
Keywords: kidney transplantation; Prediction of BK virus; Immunovirological monitoring; Associated nephropathy risk
MeSH Terms: conditions — Kidney Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — BKvirus-specific T cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Blood sample — For each patient blood (17 ml of whole blood) will be collected during a peripheral venous blood sample carried out in the the standard care at inclusion visit, M3 visit (3 months after inclusion), M6 visit (6 months after inclusion) and M12 visit (12 months after inclusion).

SUMMARY:
BKvirus associated nephropathy (BKvAN) is a major complication in kidney transplantation. Due to BKvirus (BKv) intra-graft replication, BKvAN affects nearly 10% of patients and causes graft loss in more than 50% of cases. Without current antiviral therapy, the treatment consists of minimizing immunosuppression, secondarily exposing the patient to a graft rejection risk. Impaired BKv specific T cell response plays a crucial role in the BKvAN pathophysiology. Several teams, including ours, have demonstrated a profound impairment of BKv specific T cell response during BKvAN. Immunovirological monitoring allows an individual assessment of viral reactivation risk based on the anti-viral immune response. Our group has developed the NEPHROVIR method. This non-invasive biological method allows the identification of BKvAN risk level. The aim of this work is to evaluate, by the NEPHROVIR method, the risk to develop a BKvAN with renal impairment in kidney transplant recipients with sustained BKv viremia.

The investigators propose the BK-VIR study. This is a prospective multicentric study involving 100 kidney transplant recipients with sustained BKv viremia. The aim of this work is to evaluate the NEPHROVIR method as an innovative immunovirological surveillance method for predicting the risk of BKvAN occurrence. The characterization of individual BKvAN risk level could help in the individualized follow-up and management of immunosuppression in patients. The long-term objective would be to diagnose very early, or even anticipate, the occurrence of BKvAN and to allow early readjustment of the immunosuppressive treatment.

DETAILED DESCRIPTION:
BKvirus associated nephropathy (BKvAN) is a major complication in kidney transplantation. Due to BKvirus (BKv) intra-graft replication, BKvAN affects nearly 10% of patients and causes graft loss in more than 50% of cases. Without current antiviral therapy, the treatment consists of minimizing immunosuppression, secondarily exposing the patient to a graft rejection risk. Impaired BKv specific T cell response plays a crucial role in the BKvAN pathophysiology. Several teams, including ours, have demonstrated a profound impairment of BKv specific T cell response during BKvAN. Immunovirological monitoring allows an individual assessment of viral reactivation risk based on the anti-viral immune response. Our group has developed the NEPHROVIR method. This non-invasive biological method allows the identification of BKvAN risk level. The aim of this work is to evaluate, by the NEPHROVIR method, the risk to develop a BKvAN with renal impairment in kidney transplant recipients with sustained BKv viremia.

The investigators propose the BKVIR study. This is a prospective multicentric study involving 100 kidney transplant recipients with sustained BKv viremia. Four kidney transplant centers (APHP hospitals) will participate to the study. To ensure sustained BKv viremia, only kidney transplant recipients with a confirmed plasma BKv viral load ≥ 103 copies/ml on 2 consecutive blood BKv PCR values for a duration ≥ 1 month will be eligible for the study. The investigators wish to correlate the occurrence of BKvAN with the results of the NEPHROVIR method. The primary endpoint will be the occurrence of histologically proven BKvAN associated with renal impairment within 12 months of the initial NEPHROVIR assessment. Secondary endpoints of this work are multiple, including the evaluation of the reconstitution delay of BKv specific T cell response; as well as the evaluation of the NEPHROVIR method prognosis on BKv infection and renal graft function. The expected duration of the research is 48 months. The inclusion period will be 24 months. The duration of patient follow-up will be 24 months post-inclusion. The NEPHROVIR method will be performed in the included patients at 4 distinct points: at D0 of inclusion, at 3 months, at 6 months and 12 months of inclusion. The NEPHROVIR method requires an additional and minimal collection of human body product (17 ml of whole blood) from a peripheral venous blood sample. Statistical analyses will be performed at the end of the follow-up period for all patients. All confidence intervals will be calculated at the 5% first-species risk and the results of the statistical tests will be given at the 5% two-sided threshold. The statistical analysis will be performed by the biostatisticien at the Clinical Research Unit Paris Saclay, using SAS® software or R software in the last version at the time of the analyses. The aim of this work is to evaluate the NEPHROVIR method as an innovative immunovirological surveillance method for predicting the risk of BKvAN occurrence. The characterization of individual BKvAN risk level could help in the individualized follow-up and management of immunosuppression in patients. The long-term objective would be to diagnose very early, or even anticipate, the occurrence of BKvAN and to allow early readjustment of the immunosuppressive treatment.

ELIGIBILITY:
Inclusion criteria :

* Renal transplant patients with a plasma of BK-v ≥ 103 copies/ml confirmed on 2 consecutive blood BK-V PCR values for a period of ≥ 1 month
* Men or women aged at least 18 years old - No other organ transplant except kidney transplant - Informed patient who did not object to participating in the study - Beneficiary of a social security scheme or entitled

Exclusion criteria

* Renal transplant patients with a plasma viral load of BK-v <103 copies/ml or ≥ 103 copies/ml on an isolated BK-v PCR value
* Progressive cancer apart from localized skin cancers - Occurence of acute rejection during the month prior to inclusion - Chronic progressive infectious disease (tuberculosis, replicating viral hepatitis Bor C, HIV infection), - Patient under guardianship / curatorship - Patient under State Medical Aid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Renal transplant patients with a plasma of BK-v ≥ 103 copies/ml confirmed on 2 consecutive blood BK-V PCR values for a period of ≥ 1 month aged at least 18 years old
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2021-09-02 (Actual); Primary Completion 2023-09-02 (Actual); Study Completion 2025-09-02 (Estimated)

PRIMARY OUTCOMES:
Evaluate by the NEPHROVIR method the risk of developing histologically proven BKvAN with renal impairment in kidney transplant recipients | 12 months
  The primary endpoint is the occurrence of histologically proven BKvAN with renal impairment within a maximum of 12 months after the first NEPHROVIR assessment (at inclusion: D0). Histologically proven BKvAN with renal impairment is defined as the occurrence of renal histological lesions (nuclear inclusions in tubular epithelial cells) associated with impaired renal graft function, defined as an increase in serum creatinine of more than 25% over its basal value.

SECONDARY OUTCOMES:
Assessment of the time to reconstitution of an effective anti-BK-v immune response from baseline (inclusion) at 12 months | Day 0 of inclusion, Month 3, Month 6 and Month 12 post-inclusion
  This assessment will be based on the kinetics of evolution between repeated measurements of the NEPHROVIR method (at Day 0 of inclusion, Month 3, Month 6 and Month 12 post-inclusion).
Assessment of the prognostic character of NEPHROVIR on BKv infection from baseline (inclusion) at 12 months | Day 0 of inclusion, Month 3, Month 6 and Month 12 post-inclusion
  This assessment will be based on the kinetics of the evolution between repeated NEPHROVIR measurements (at Day 0 of inclusion, Month 3, Month 6 and Month 12 post-inclusion) and repeated BKv viral load (assessed by PCR at D0 of inclusion and then every 3, 6, and 12 months).
Assessment of the prognostic character of NEPHROVIR on kidney graft function from baseline (inclusion) at 24 months | Day 0 of inclusion, Month 3, Month 6, Month 12 and Month 24 post-inclusion
  This assessment will be based on the kinetics of the evolution between repeated NEPHROVIR measurements (at Day 0 of inclusion, Month 3, Month 6 and Month 12 post-inclusion) and repeated plasma creatinine measurements of patients on the day of inclusion in the study and at 3, 6, 12 and 24 months post-inclusion.
Assessment of the prognostic character of NEPHROVIR on kidney graft allorejection risk from baseline (inclusion) at 12 months | Day 0 of inclusion, Month 3, Month 6 and Month 12 post-inclusion
  This evaluation will be based on the kinetics of the evolution between repeated measurements of NEPHROVIR (at Day 0 of inclusion, Month 3, Month 6 and Month 12 post-inclusion) and the occurrence of graft rejection or graft lost.

CONTACTS AND LOCATIONS:
Overall Officials: Antoine DURRBACH, profesor, Principal Investigator — Henri Mondor University Hospital
Locations (5):
- France (5):
  - Henri Mondor Hospital (001), Créteil
  - Saint Louis Hospital (003), Paris
  - La Pitié Salpêtrière Hospital (004), Paris
  - Necker Hospital (005), Paris
  - Foch Hospital (002), Suresnes

IPD SHARING:
Plan to Share IPD: No